CLINICAL TRIAL: NCT06995924
Title: A Pilot Trial to Evaluate the Effectiveness of Navigation, Interactive Web Education, or the Combination of Both to Promote Guideline-Concordant Colorectal Cancer Surveillance Care
Brief Title: Improving Uptake of Surveillance in Colorectal Cancer Survivors Through Navigation and Web Education
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1125283; NCI-2025-03304 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20875 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-08

CONDITIONS: Stage I Colorectal Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (navigation) (Experimental): Patients at the Virginia Mason clinic location receive access to navigation services, in person, via telephone or via electronic conferencing platform, including education on surveillance care, reminders to complete care and assistance in scheduling surveillance, within 3 months of standard of care surgical resection.
  Interventions: Other: Electronic Health Record Review; Behavioral: Patient Navigation; Other: Survey Administration
- Arm B (CTAC) (Experimental): Patients at the Fred Hutch (South Lake Union) clinic location receive access to the online CTAC intervention, which includes self-directed, interactive education about surveillance and a checklist of care, within 3 months of standard of care surgical resection.
  Interventions: Other: Educational Intervention; Other: Electronic Health Record Review; Other: Internet-Based Intervention; Other: Survey Administration
- Arm C (navigation and CTAC) (Experimental): Patients at the Fred Hutch (Overlake) clinic location receive access to navigation services, in person, via telephone or via electronic conferencing platform, including education on surveillance care, reminders to complete care and assistance in scheduling surveillance, and access to the online CTAC intervention, which includes self-directed, interactive education about surveillance and a checklist of care, within 3 months of standard of care surgical resection.
  Interventions: Other: Educational Intervention; Other: Electronic Health Record Review; Other: Internet-Based Intervention; Behavioral: Patient Navigation; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Complete self-directed interactive education
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm B (CTAC); Arm C (navigation and CTAC)
Other: Electronic Health Record Review — Ancillary studies
Other: Internet-Based Intervention — Receive access to CTAC
  Arms: Arm B (CTAC); Arm C (navigation and CTAC)
Behavioral: Patient Navigation — Receive patient navigation services
  Other Names: Patient Navigator Program
  Arms: Arm A (navigation); Arm C (navigation and CTAC)
Other: Survey Administration — Ancillary studies

SUMMARY:
This pilot clinical trial looks at whether patient navigation services, an interactive web education intervention, called Current Together After Cancer (CTAC), or both navigation and CTAC works to improve the uptake of surveillance in patients with stage I-III colorectal cancer (CRC). Post-treatment surveillance is critical to detect recurrence early, yet many CRC survivors do not receive recommended surveillance care. Surveillance is a complex process that includes laboratory tests, cross-sectional imaging, and endoscopic procedures. Patient navigation services, interactive web education, or a combination of both may improve surveillance care for patients with stage I-III colorectal cancer.

DETAILED DESCRIPTION:
OUTLINE:

Patients are assigned to 1 of 3 arms based on the clinic location they receive cancer care at.

ARM A (VIRGINIA MASON): Patients receive access to navigation services, including education on surveillance care, reminders to complete care and assistance in scheduling surveillance, within 3 months of standard of care surgical resection for stage I-III CRC.

ARM B (FRED HUTCH [SOUTH LAKE UNION]): Patients receive access to the CTAC intervention, which includes self-directed, interactive web-based education about surveillance and a checklist of care, within 3 months of standard of care surgical resection for stage I-III CRC.

ARM C (FRED HUTCH [OVERLAKE]): Patients receive access to navigation services, including education on surveillance care, reminders to complete care and assistance in scheduling surveillance, and access to the CTAC intervention, which includes self-directed, interactive web-based education about surveillance and a checklist of care, within 3 months of standard of care surgical resection for stage I-III CRC.

Patients are followed up at 3 and 9 months post study-enrollment and 12-18 months after surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 due to disease and clinic population
* Stage I-III CRC survivor within 3 months post-surgical resection
* Being seen at a participating clinic
* Ability to understand and complete surveys in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Completion of colonoscopy (stage I colorectal carcinoma patients) | Up to 18 months post-surgical resection
Completing any colonoscopy, carcinoembryonic antigen tumor marker (CEA), and cross-sectional imaging (stage II-III colorectal carcinoma patients) | Up to 18 months post-surgical resection
  Will compare rates of surveillance care completion 1-year (up to 18 months accounting for delays that may be due to inability accessing endoscopy) post-surgical resection across groups using chi-square tests. Will use a multivariable logistic regression model to test for factors that may be associated with increased or decreased surveillance care including patient-level demographic factors (e.g., age, sex, etc.) and available clinic-level factors (e.g., clinic size, etc.).

SECONDARY OUTCOMES:
Knowledge of colorectal cancer (CRC) surveillance | At baseline, 3 and 9 months post enrollment
  Knowledge will be assessed using a previously validated 5-item scale. Responses will be graded on a scale of 0 to 5 with higher scores representing higher knowledge; scores can also be dichotomized into high and low knowledge.
Self-efficacy to complete CRC surveillance | At baseline, 3 and 9 months post enrollment
  Will be measured using 7-items on a 5-point Likert scale ("strongly disagree" to "strongly agree"). Responses will be averaged with higher scores indicating greater self-efficacy.
Acceptability of the intervention | At 3 and 9 months post enrollment
  Assessed using Acceptability of the Intervention Measure. Will calculate and compare mean scores between individual participants and exposure group using student's t-test.
Intervention appropriateness | At 3 and 9 months post enrollment
  Assessed using Intervention Appropriateness Measure (IAM). Will calculate and compare mean scores between individual participants and exposure group using student's t-test.
Feasibility of the intervention | At 3 and 9 months post enrollment
  Assessed using Feasibility of Intervention Measure (FIM) scores. Will calculate and compare mean scores between individual participants and exposure group using student's t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel B. Issaka, MD, MAS, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No